CLINICAL TRIAL: NCT03563638
Title: Maternal Serum Pentraxin 3 in Early Pregnancy to Predict Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Quxiaoxian
Record Dates: First submitted 2018-05-26; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Pregnancy Complications Affecting Fetus (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GDM group: Women with maternal age ≥ 18 years, singleton pregnancy, primipara, no smoking, confirmed gestation≤20 weeks and spontaneous conception were invited to participate in the study,and excluded if they had multiple pregnancy, pre-gestational diabetes mellitus, hypertensive disorders, preterm delivery, cardiovascular disease, immunological disease, glucocorticoid therapy, or other severe illness,and fetal abnormalities occurred during pregnancy were also excluded from the study.GDM was verified on the 75gOGTT at 24-28 gestational weeks.The diagnosis of GDM is made when any of the following plasma glucose values are met or exceeded: FPG≥5.1 mmol/L and/or 1h-PG ≥10.0 mmol/L and/or 2h-PG ≥8.5 mmol/ L.
  Interventions: Diagnostic Test: 75gOGTT
- NGT group: Women with maternal age ≥ 18 years, singleton pregnancy, primipara, no smoking, confirmed gestation≤20 weeks and spontaneous conception were invited to participate in the study. Women were excluded if they had multiple pregnancy, pre-gestational diabetes mellitus (PGDM), hypertensive disorders, preterm delivery, cardiovascular disease, immunological disease, glucocorticoid therapy, or other severe illness. if there were fetal abnormalities including chromosomally abnormal fetuses and/or structural defects and fetal growth restriction occurred during pregnancy were also excluded from the study.GDM was verified on the 75gOGTT at 24-28 gestational weeks.those who not met the criteria were the NCT group.
  Interventions: Diagnostic Test: 75gOGTT

INTERVENTIONS:
Diagnostic Test: 75gOGTT — oral glucose tolerance test (OGTT) was conducted on all participants between the 24th and 28th gestation weeks.The diagnosis of GDM is made when any of the following plasma glucose values are met or exceeded: FPG≥5.1 mmol/L and/or 1h-PG ≥10.0 mmol/L and/or 2h-PG ≥8.5 mmol/ L.

SUMMARY:
To investigate the association of maternal serum concentrations of pentraxin 3 in early pregnancy with gestational diabetes mellitus and to explore its potential value in the prediction of GDM.

DETAILED DESCRIPTION:
We recruited all pregnant women for the first checkup in our hospital . Maternal fasting serum PTX3 levels, fasting plasma glucose and fasting insulin and other factors were measured. Oral glucose tolerance test (OGTT) was performed at 24-28 weeks in all participants. According to the occurrence of GDM, subjects were divided into two groups: GDM group and normal glucose tolerance (NGT) group.

ELIGIBILITY:
Inclusion Criteria:

* Women with maternal age ≥ 18 years, singleton pregnancy, primipara, no smoking, confirmed gestation≤20 weeks and spontaneous conception were invited to participate in the study.

Exclusion Criteria:

* Women were excluded if they had multiple pregnancy, pre-gestational diabetes mellitus (PGDM), hypertensive disorders, preterm delivery, cardiovascular disease, immunological disease, glucocorticoid therapy, or other severe illness. In addition, women who were suffering from fetal abnormalities including chromosomally abnormal fetuses and/or structural defects and fetal growth restriction occurred during pregnancy were also excluded from the study.

Ages: 27 Years to 33 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: chinese women with maternal age ≥ 18 years, singleton pregnancy, primipara, no smoking, confirmed gestation≤20 weeks and spontaneous conception
Sampling Method: Probability Sample
Enrollment: 824 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Serum PTX3 levels in early pregnancy | 2015.10.01-2015.11.31
  Serum PTX3 levels in early pregnancy